CLINICAL TRIAL: NCT01660802
Title: Safety and Efficacy Study of Dexamethasone in the Treatment of Patients With Macular Edema Following Retinal Vein Occlusion (RVO)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 206207-020
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Macular Edema
MeSH Terms: conditions — Macular Edema | interventions — Dexamethasone; Calcium Dobesilate; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 700 μg Dexamethasone (Experimental): 700 μg Dexamethasone intravitreal injection in the study eye on Day 1.
  Interventions: Drug: 700 μg Dexamethasone
- Sham (Sham Comparator): Sham administered in the study eye on Day 1.
  Interventions: Drug: 700 μg Dexamethasone; Other: Sham

INTERVENTIONS:
Drug: 700 μg Dexamethasone — 700 μg Dexamethasone intravitreal injection in the study eye on Day 1.
  Other Names: Ozurdex®
Other: Sham — Sham administered in the study eye on Day 1.
  Arms: Sham

SUMMARY:
This study will assess the safety and efficacy of 700 μg dexamethasone Posterior Segment Drug Delivery System (DEX PS DDS) Applicator System in patients with macular edema in a 6 month double-blind period versus sham followed by a 2 month open label period.

ELIGIBILITY:
Inclusion Criteria:

-Presence of macular edema defined as macular thickening involving the center of the macula due to branch retinal vein occlusion (BRVO) or central retinal vein occlusion (CRVO)

Exclusion Criteria:

* History of glaucoma, ocular hypertension or optic nerve head change
* Any active bacterial, viral, parasitic, or fungal infections in either eye
* Eye surgery, including cataract surgery, and/or laser of any type in the study eye within 3 months prior to study start
* History of use of intravitreal steroids or any intravitreal injectable drug in the study eye within 3 months prior to study start
* Use of oral, intravenous, intramuscular, epidural, rectal, or extensive dermal steroids within 1 month prior to study start
* Use of immunosuppressants, immunomodulators, antimetabolites, and/or alkylating agents within 3 months prior to study start
* Use of topical ophthalmic corticosticosteroids within 2 weeks of study start

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2012-09-04 (Actual); Primary Completion 2014-03-31 (Actual); Study Completion 2014-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Beijing, China

REFERENCES:
- [Background] Li X, Wang N, Liang X, Xu G, Li XY, Jiao J, Lou J, Hashad Y; China Ozurdex in RVO Study Group. Safety and efficacy of dexamethasone intravitreal implant for treatment of macular edema secondary to retinal vein occlusion in Chinese patients: randomized, sham-controlled, multicenter study. Graefes Arch Clin Exp Ophthalmol. 2018 Jan;256(1):59-69. doi: 10.1007/s00417-017-3831-6. Epub 2017 Nov 8. PMID 29119239

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 700 μg Dexamethasone | Sham
Started | 130 | 132
Completed | 126 | 121
Not Completed | 4 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 700 μg Dexamethasone | Sham | Total
Number analyzed (Participants) | 130 | 132 | 262
Age, Customized [Number; unit: Participants]
  <45 years | 18 | 25 | 43
  45 to 65 years | 94 | 86 | 180
  > 65 years | 18 | 21 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 76 | 136
  Male | 70 | 56 | 126

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With 15 or More Letter Improvement in Best Corrected Visual Acuity (BCVA) in the Study Eye
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. The numbers of patients with at least a 15 or more letter improvement in BCVA in the study eye are presented.
Time Frame: Baseline, 6 Months
Population: Modified Intent-to-Treat: all randomized and treated patients
Measure: Number; unit: Patients
Arm/Group | 700 μg Dexamethasone | Sham
Number analyzed (Participants) | 129 | 130
Patients | 60 | 31

2. Secondary Outcome: Average Change From Baseline in BCVA in the Study Eye
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The average BCVA is calculated across study visits for each patient. A positive number change from baseline indicates an improvement and a negative number change from baseline indicates a worsening.
Time Frame: Baseline, 6 Months
Population: Modified Intent-to-Treat: all randomized and treated patients
Measure: Mean (Standard Deviation); unit: Letters Read Correctly
Arm/Group | 700 μg Dexamethasone | Sham
Number analyzed (Participants) | 129 | 130
Letters Read Correctly
  Baseline | 52.6 (10.79) | 53.1 (10.47)
  Average Change from Baseline Over 6 Months | 6.6 (8.98) | 2.5 (9.98)

3. Secondary Outcome: Change From Baseline in BCVA in the Study Eye
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. A decrease in the number of letters read correctly (negative number) means that vision has worsened.
Time Frame: Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6
Population: Modified Intent-to-Treat: all randomized and treated patients
Measure: Mean (Standard Deviation); unit: Letters Read Correctly
Arm/Group | 700 μg Dexamethasone | Sham
Number analyzed (Participants) | 129 | 130
Letters Read Correctly
  Baseline | 52.6 (10.79) | 53.1 (10.47)
  Change from Baseline at Month 1 | 9.1 (8.45) | 2.0 (9.28)
  Change from Baseline at Month 2 | 10.6 (10.36) | 1.7 (12.29)
  Change from Baseline at Month 3 | 7.7 (12.66) | 1.8 (12.98)
  Change from Baseline at Month 4 | 5.2 (12.79) | 3.3 (12.32)
  Change from Baseline at Month 5 | 4.4 (13.28) | 3.3 (13.04)
  Change from Baseline at Month 6 | 3.2 (15.34) | 4.0 (13.73)

4. Secondary Outcome: Percentage of Patients With BCVA Improvement of ≥15 Letters From Baseline in the Study Eye
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly indicates improvement and a decrease in the number of letters read correctly indicates a worsening.
Time Frame: Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6
Population: Modified Intent-to-Treat: all randomized and treated patients
Measure: Number; unit: Percentage of Patients
Arm/Group | 700 μg Dexamethasone | Sham
Number analyzed (Participants) | 129 | 130
Percentage of Patients
  Month 1 | 28.7 | 5.4
  Month 2 | 34.9 | 11.5
  Month 3 | 33.3 | 13.1
  Month 4 | 23.3 | 14.6
  Month 5 | 22.5 | 22.3
  Month 6 | 23.3 | 20.8

ADVERSE EVENTS:
Description: The Safety Population included all treated patients and was used to assess adverse events (AEs) and serious adverse events (SAEs). Treatment emergent adverse events (TEAE) are reported and include all AEs and SAEs that began or worsened after study treatment.
Arm/Group | 700 μg Dexamethasone | Sham
Serious Adverse Events (participants affected / at risk) | 1/129 | 2/130
Other Adverse Events (participants affected / at risk) | 69/129 | 15/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 700 μg Dexamethasone (N=129) | Sham (N=130)
Atrioventricular Block (Cardiac disorders) | 1 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 0 | 1
Vitreous Haemorrhage (Eye disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 700 μg Dexamethasone (N=129) | Sham (N=130)
Conjunctival Haemorrhage (Eye disorders) | 24 | 5
Conjunctival Hyperaemia (Eye disorders) | 17 | 6
Intraocular Pressure Increased (Investigations) | 38 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for at least 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.